CLINICAL TRIAL: NCT05454501
Title: The Effects of Telerehabilitation and Exercise Training on Physical Activity, Exercise Capacity, Muscle Strength and Quality of Life in Pediatric Arrhythmia Patients With Pacemakers
Brief Title: The Effects of Telerehabilitation and Exercise Training in Pediatric Arrhythmia Patients With Pacemakers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sena Teber, Lecturer, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E-22481095-020-1222
Record Dates: First submitted 2022-05-31; First posted 2022-07-12 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-05

CONDITIONS: Congenital Heart Disease
Keywords: pacemaker; physical activity; exercise; live videoconferencing; quality of life; cardiac rehabilitation
MeSH Terms: conditions — Heart Defects, Congenital; Motor Activity | interventions — Exercise; Patient Education as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Training (Active Comparator): 8-week real-time online exercise training will be provided. The content of the training will be aerobic based exercises, strength and flexibility exercises with warm up and cool down phases.
  Interventions: Other: Exercise Training
- Patient Education (Active Comparator): Patients will be given face-to-face education about their disease, the importance of physical activity and how to do it safely. They will be followed up with information leaflets and weekly phone calls.
  Interventions: Other: Patient Education

INTERVENTIONS:
Other: Exercise Training — For eight weeks, they will receive real-time online exercise training for 30 minutes, three days a week, with a peer group of 5-6 people. Before starting the exercise, physical activity will be monitored for seven days.
  Arms: Exercise Training
Other: Patient Education — After the first face-to-face evaluation session, these patients and their families will receive a 1-hour patient education program specific to the disease and exercise. Information brochures containing physical activity and exercise recommendations will be given. They will be followed up with weekly phone calls throughout the study period. At the end of 8 weeks, the second evaluation interview will be held. Afterward, the patients in the control group will be able to participate in the online exercise training program if they request it.
  Arms: Patient Education

SUMMARY:
There is no study evaluating online exercise training and results in children with pacemakers. This study investigates the effects of group exercise training performed via computer online videoconferencing in pediatric arrhythmia patients with pacemakers. Pediatric arrhythmia patients aged 6-18 years with a pacemaker, stable clinically, and living with at least one parent or caregiver who can support them at home will be included in the study. Eligible patients will be randomly divided into two groups. After the face-to-face evaluation session, those in the intervention group will receive real-time online exercise training for 30 minutes, three days a week, with a peer group of 5-6 people for eight weeks. Physical activity will be monitored for seven days before starting the exercise and seven days after the training is completed. After the first face-to-face evaluation session, patients in the control group and their families will receive a 1-hour disease- and exercise-specific patient education program. Information brochures containing physical activity and exercise recommendations will be given. They will be followed up with weekly phone calls throughout the study period.

DETAILED DESCRIPTION:
It is known that physical activity and exercise have long-term beneficial effects on preventing atherosclerotic cardiovascular diseases, dyslipidemia, obesity, hypertension, osteoporosis, and type 2 diabetes, frequently seen in sedentary individuals. Various exercise training programs are safe and feasible and improve functional outcome measures in this patient population. Walking distance, peak oxygen consumption, and increased physical activity were observed in these patients with exercise training. Increasing physical activity in children is also associated with gross motor performance development and positive emotional, social, and intellectual development. The probability of being a sedentary adult was very low in congenital heart patients who do sports from an early age. Universal reports drew attention to the importance of exercise and physical activities in children with heart disease and stated that they should be encouraged. Paradoxically, only a minority of children with heart disease receive physical activity counseling. Children with pacemakers have similar potential to improve their physical fitness through physical activity as their healthy peers. However, children often experience an uncertainty about what physical activities should be recommended and how the intensity of exercise should be, and they are brought up with overprotective attitudes. This encourages children to inactivity and causes them to feel inadequacy and fear. In addition, patient and family concerns about the particular vulnerability of children with pacemakers; may exacerbate social isolation and physical inactivity more than the general population. .

Exercise training may be the most crucial strategy to improve functional capacity, increase physical activity and reduce the risk of future cardiovascular events. Although consensus reports indicated that exercise should be encouraged and performed regularly in these patients, it is not a common practice. Among the possible reasons; are logistical problems, costs, and parental concern about adverse events. There is a need to evaluate the effects of rehabilitation programs that can connect safely and inexpensively with these patients, including those living geographically far from rehabilitation centers. Home-based exercise approaches can be preferred as a safe, feasible, and beneficial alternative to supervised cardiac rehabilitation for all age groups with congenital hearth disease. The effectiveness of online exercise programs provided or supported through the Internet and related technologies is safe for children to participate in and improve compliance.

The potential of online exercise programs in children with congenital hearth disease remains largely unexplored. Although no study evaluates exercise training and results in pediatric arrhythmia patients with pacemakers, the subject is open to research.

ELIGIBILITY:
Inclusion Criteria:

* stable clinical condition (having a medical examination in the last three months, including an ECG and an echocardiogram),
* living with at least one parent or caregiver who can support them at home

Exclusion Criteria:

* To have any neurological, advanced orthopedic problems, any other systemic disease or acute infection,
* To use anticoagulant drugs,
* To have Down syndrome,
* Cannot cooperate with the video conference system and measurements

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Number of steps | for 7 consecutive days before and after training days. Change from baseline to 8 weeks.
  It will be evaluated with an activity tracker
Perceived effort, maximum workload and heart rate reserve | A week before before starting the training and after 8 weeks training. Change from baseline to 8 weeks.
  Cardiorespiratory capacity will be evaluated with an effort test with a treadmill. The modified Bruce protocol will be used as the treadmill protocol.
6 Minute Walk Test (6MWT) Walking Distance | A week before before starting the training and after 8 weeks training. Change from baseline to 8 weeks.
  Functional exercise capacity will be assessed with the 6 Minute Walk Test. Pre-test heart rate, blood pressure, saturation values will be evaluated during and after the test.

SECONDARY OUTCOMES:
peripheral muscle strength | A week before before starting the training and after 8 weeks training. Change from baseline to 8 weeks.
  hand dynamometer
health related quality of life | A week before before starting the training and after 8 weeks training. Change from baseline to 8 weeks.
  PedsQL self-reported quality of life scale

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit and Hacettepe University Faculty of Medicine, Department of Pediatrics, Department of Pediatric Cardiology, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided